CLINICAL TRIAL: NCT03654521
Title: Fetal Interventricular Septum Thickness and Maternal Gestational Diabetes Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yaniv Zipori MD, Principal Investigator, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0580-17-RMB
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes group (Active Comparator): Women with gestational or pre-gestational diabetes mellitus.
  Interventions: Diagnostic Test: Fetal interventricular septum thickness
- Control group (Active Comparator): Women without gestational or pre-gestational diabetes mellitus.
  Interventions: Diagnostic Test: Fetal interventricular septum thickness

INTERVENTIONS:
Diagnostic Test: Fetal interventricular septum thickness — Two-dimensional ultrasound fetal cardiac imaging test

SUMMARY:
Glucose intolerance and gestational diabetes are common complications of pregnancy. Their prevalence varies worldwide secondary to differences in screening practices (one-step versus two-step approach) and population characteristics (increased maternal age, body mass index, ethnicity). Gestational diabetes mellitus is associated with increased incidence of macrosomia, operative vaginal delivery, shoulder dystocia, cesarean delivery, metabolic complications in the newborn and long-term risk of developing type II diabetes mellitus (HAPO 2008).

Early diagnosis and management of gestational diabetes mellitus, including dietary advice and insulin, improves maternal and fetal outcomes (Crowther 2005, Hartling 2013). Various strategies have been tested prenatally to detect those fetuses that might be adversely affected by gestational diabetes mellitus. For instance, the abdominal circumference measurement during routine fetal biometry was used successfully to identify pregnancies with a higher risk of fetal macrosomia (Schaefer-Graf 2003, De Reu 2008, Rosati 2010). In recent years, the fetal interventricular septum thickness, as detected by two-dimensional ultrasound, was shown to be significantly thicker in the presence of gestational diabetes mellitus, independently of maternal glycemic control, when compared to pregnancies with no gestational diabetes mellitus (Ren 2011, Garg 2014).

Current guidelines focus on normalisation of maternal blood glucose concentration. Thus far no study has addressed whether measurement of the fetal interventricular septum thickness can predict adverse pregnancy outcome in euglycemic women with gestational diabetes mellitus.

DETAILED DESCRIPTION:
Rational for the study If fetal interventricular septum hypertrophy in pregnancies with gestational diabetes mellitus appears prior to either fetal abdominal circumference measurement > 90th percentile or the abnormal maternal glucose levels, then future management of women with gestational diabetes mellitus might be targeted earlier at these pregnancies to ensure a more favorable outcome.

Objective To determine the thickness of fetal interventricular septum in women with and without gestational diabetes mellitus and correlates it with perinatal outcome.

Methods Study design This is a prospective study at Rambam Health Care Campus. Inclusion / Exclusion criteria

1. Inclusion Study group - women between 24 - 34 weeks' gestation who were diagnosed with gestational diabetes mellitus or known with type I or type II diabetes mellitus.

   Control group - women between 24 - 34 weeks' gestation who do not have diabetes.
2. Exclusion (that might affect directly or indirectly the fetal cardiac function) - women who did not complete a glucose challenge test, smoking, underlying cardiac or respiratory illness, fetal growth restriction, medicated hypertension disorder of pregnancy, multiple pregnancy, use of steroids for lung maturation in the current pregnancy and known major congenital anomalies.

Study population Women who meet the above inclusion criteria will be asked to participate in the study, and will be asked to provide a written informed consent. Both groups, the study and control group, will be recruited when attending their routine prenatal care in the prenatal clinics at Rambam Health Care Campus. Eligible woman will undergo ultrasound examination as they would normally do in each visit. This study, under no circumstances, will alter the participants routine care.

Data Collection

1. Maternal and fetal characteristics Data related to the fetomaternal antenatal, intrapartum and postpartum course will be recorded prospectively (Appendix 1).
2. Ultrasound assessment Basic transabdominal two-dimensional ultrasound examination using B-mode (either Samsung or Voluson E8), will be carried out first to assess fetal growth and well-being. This is to be continued with a more detailed ultrasound, with a specific focus on the fetal interventricular septum. The entire length of the study, dependent on fetal lie, is expected to take around 15 min. The results of the assessment of fetal growth and well-being will be provided to the patient.

The measurement of the fetal interventricular septum will be as follow (Figure 1 below); maternal suspended respiration, without fetal movement or breathing, level of the 4-chamber view with adequate magnification of the fetal heart (50% of the screen), midpoint of interventricular septum with cine loop to end-diastolic (maximum ventricular filling), and average of 3 measurements (Ren 2011, Garg 2014).

ELIGIBILITY:
Inclusion Criteria:

* Study group - women between 24 - 34 weeks' gestation who were diagnosed with gestational diabetes mellitus or known with type I or type II diabetes mellitus.

Control group - women between 24 - 34 weeks' gestation who do not have diabetes.

Exclusion Criteria:

* women who did not complete a glucose challenge test, smoking, underlying cardiac or respiratory illness, fetal growth restriction, medicated hypertension disorder of pregnancy, multiple pregnancy, use of steroids for lung maturation in the current pregnancy and known major congenital anomalies.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 500 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Fetal interventricular septum thickness | Between 24-34 weeks of gestation.
  Differences in fetal interventricular septum thickness in both women with gestational or pre-gestational diabetes mellitus and women without gestational or pre-gestational diabetes mellitus.

CONTACTS AND LOCATIONS:
Overall Officials: Yaniv Zipori, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel